CLINICAL TRIAL: NCT05766488
Title: Assessing Continuous Glucose Monitor Use in Underserved Primary Care Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Great Plains IDeA-CTR (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0314-22-FB
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Glucose Self-Monitoring

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups and receive either the treatment intervention, continuous glucose monitor (CGM), or standard of care intervention ,traditional glucometer, upon enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Continuous Glucose Monitoring (Experimental): Participants will use a Freestyle Libre 2 monitoring device for 6 months to track blood glucose levels.
  Interventions: Device: Continuous Glucose Monitor (CGM)
- Traditional Glucometer Arm (Active Comparator): Participants will use a traditional glucose monitoring device (glucometer) to self-monitor their blood glucose for 6 months to track blood glucose levels.
  Interventions: Device: Self-monitoring Blood Glucose (SMBG)

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — A Freestyle Libre 2 continuous glucose monitor (CGM) will be provided in the experimental arm of this study for 6 months.
  Other Names: Flash-glucose Monitor
  Arms: Continuous Glucose Monitoring
Device: Self-monitoring Blood Glucose (SMBG) — A traditional glucometer device will be assigned in the active comparitor arm of this study for 6 months.
  Other Names: Traditional glucometer
  Arms: Traditional Glucometer Arm

SUMMARY:
Continuous glucose monitoring (CGM) has demonstrated improved outcomes in both type 1 and type 2 diabetes populations in comparison to traditional methods; however, these devices have not been well studied in underserved adult patients (e.g., low-income, uninsured) who may face additional barriers to monitoring. Furthermore, there is limited data exploring long-term (3- to 6- month) health care team-based management of these devices in the primary care setting. The purpose of this study is to further understand the benefits and barriers associated with CGM use in underserved populations with type 2 diabetes and improve their overall diabetes care.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) has demonstrated improved outcomes in both type 1 and type 2 diabetes populations in comparison to traditional methods; however, these devices have not been well studied in underserved adult patients (e.g., low-income, uninsured) who may face additional barriers to monitoring. Furthermore, there is limited data exploring long-term (3- to 6- month) health care team-based management of these devices in the primary care setting. This study will evaluate the perceived and experienced benefits and barriers of continuous glucose monitor (CGM) and traditional glucometer use and identify diabetes related outcomes associated with CGM use relative to usual care with self-monitoring of blood glucose (SMBG) in an underserved population.

Eligible adult (>=19 years of age) patients at participating clinics with type 2 diabetes, A1c >=9%, and concomitant insulin therapy and/or using two or more diabetes medications will be randomly enrolled to one of two groups: Freestyle Libre 2 CGM or traditional glucometer. Pre- and post-surveys will be used to evaluate perceived and experienced benefits and barriers to CGM use and diabetes-related outcomes will be compared between the groups using face-to-face, telephonic, and/or digital avenues. The latter aim will replicate current processes of team-based diabetes care which is blood glucose management from a pharmacist under collaborative practice with the primary care physician. Follow-up will also replicate these clinic processes throughout the 6-month period, including telephone calls and monthly in-clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* A1c >9% at recruitment
* On/initiating insulin or on two or more diabetes medications

Exclusion Criteria:

* Current use of an insulin pump
* On dialysis
* Pregnant
* Implanted medical device (e.g., pace-maker, defibrillator)
* Intellectual or physical disabilities that may interfere with ability to properly use the Continuous Glucose Monitor (CGM)
* Able to read English

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (Hemoglobin A1c) | Baseline, 3 months, and 6 months.
  Glycemic control will be assessed by measuring hemoglobin A1c at baseline, 3 months, and 6 months. Values will be evaluated as a continuous variable and categorized as <7.0% vs >7.0% to <9.0% and >9.0%. Comparisons of the proportions of participants achieving a minimum of 1 point drop in hemoglobin A1c will be made between study arms.

SECONDARY OUTCOMES:
Hypoglycemia | 6 months
  Continuous glucose monitor (CGM) and glucometer blood glucose data will be evaluated to determine number and percentage of hypoglycemic readings (i.e., <70 mg/dL). For CGM data, % time within target range, % time below specific thresholds for hypoglycemia) will be captured and described.
Hyperglycemia | 6 months
  Continuous glucose monitor (CGM) and glucometer blood glucose data will be evaluated to determine percentage of hyperglycemic values (i.e., >180 mg/dl) experienced. For CGM data, % time within target range, % time below specific thresholds for hypoglycemia) will be captured and described.
Blood Glucose Capture Rate | 6 months
  Number of days without any blood glucose recordings will be captured as a percentage over the study period.
Perceived or Experienced Benefits and Barriers to Device Use | Baseline and 6 months
  A pre- and post-survey will be provided to all participants to qualitatively identify benefits and barriers to access and use of their assigned device and willingness to continue CGM use (follow-up survey).

CONTACTS AND LOCATIONS:
Overall Officials: Drew C Prescott, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- Nebraska Medicine, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No